CLINICAL TRIAL: NCT03961958
Title: Relationship Between Hemodynamic Changes and Propofol Pharmacokinetic Variation During Anesthesia Induction and Knee-chest Positioning in Propofol TCI Guided Anesthesia
Brief Title: Hemodynamic Changes and Propofol Pharmacokinetic Variation During Anesthesia Induction and Knee-chest Positioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Daniela Chalo, Principal Investigator, University of Salamanca
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: USalamanca
Record Dates: First submitted 2019-05-11; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Hemodynamic Instability; Anesthesia; Surgery
Keywords: Hemodynamics; Knee-Chest Position; Propofol; Anesthesia, General; Anesthetics, Intravenous; pharmacokinetics

STUDY DESIGN:
Intervention Model Description: In phase 1, target-controlled infusion propofol anesthesia was adjusted to maintain BIS 40 to 60.
  In phase 2, there were 2 planned reductions in propofol target concentration: (1) immediately after loss of consciousness - reduction calculated using a predefined formula, and (2) before positioning - reduction equal to the average percentage decrease in CO after knee-chest position in phase 1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No protocolled propofol reduction (No Intervention): In phase 1, target-controlled infusion propofol anesthesia was adjusted to maintain BIS 40 to 60.
- Two protocolled propofol reductions (Experimental): In phase 2, there were 2 planned reductions in propofol target concentration: (1) immediately after loss of consciousness-reduction calculated using a predefined formula, and (2) before positioning-reduction equal to the average percentage decrease in CO after knee-chest position in phase
  Interventions: Drug: Propofol reduction

INTERVENTIONS:
Drug: Propofol reduction — Reduction of propofol target concentration
  Arms: Two protocolled propofol reductions

SUMMARY:
Induction of anesthesia and the knee-chest position are associated with hemodynamic changes that may impact patient outcomes.

Changes from baseline in cardiac output and other hemodynamic variables following induction of anesthesia and knee-chest positioning were compared. Propofol plasma concentrations were also measured after induction of anesthesia and after the knee-chest position.

The aim of this study was to assess whether planned reductions in target-controlled infusion propofol concentrations attenuate the hemodynamic changes associated with anesthesia induction and knee-chest position.

The secondary aim was to quantify the variation in propofol measured plasma concentrations (Cm), both after induction and after KC positioning, and correlate them with predicted concentrations (Cp) by the Schnider Pk model.

DETAILED DESCRIPTION:
A total of 20 patients scheduled for elective lumbar spinal surgery in the knee-chest position were included. In addition to standard anesthesia monitoring, bispectral index and noninvasive cardiac output monitoring were undertaken. The study was carried out in 2 parts. In phase 1, target-controlled infusion propofol anesthesia was adjusted to maintain BIS 40 to 60. In phase 2, there were 2 planned reductions in propofol target concentration: (1) immediately after loss of consciousness: reduction calculated using a predefined formula, and (2) before positioning: reduction equal to the average percentage decrease in CO after knee-chest position in phase 1.

ELIGIBILITY:
Inclusion Criteria:

• Lumbar spinal condition for surgical treatment in knee-chest position

Exclusion Criteria:

* Severe ischemic heart disease
* Congestive heart failure
* Atrial fibrillation or flutter
* Body mass index > 35 kg/m2
* Glasgow Coma Scale < 15
* Dementia disease
* History of drug abuse or addiction
* Consumption of opioid medication
* Pre-operative administration of midazolam

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Hemodynamic changes | Baseline (moment 0), 10 minutes after induction of anesthesia (moment 1), 10 minutes after knee-chest positioning (moment 2)
  Changes from baseline in cardiac output and comparison of the changes between both groups.

SECONDARY OUTCOMES:
Pharmacokinetic changes | Baseline (moment 0), 10 minutes after induction of anesthesia (moment 1), 10 minutes after knee-chest positioning (moment 2)
  Correlation between propofol measured plasma concentrations and predicted plasma concentrations (Cp) by the Schnider Pk model.

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo S Sanchez, PhD, Study Director — University of Salamanca, Faculty of Medicine
Locations (1):
- Centro Hospitalar do Porto, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, CSR
Time Frame: starting 6 months from publication, for 1 year
Access Criteria: everyone who asks for access after the explanation